CLINICAL TRIAL: NCT05186181
Title: Endovascular Repair of Stanford B-type Thoracic Aortic Dissection With Insufficient Proximal Landing Zone by Left Subclavian Artery in Situ Stent Graft Puncture and Fenestration: A Prospective, Single-arm, Observational Clinical Trial.
Brief Title: Endovascular Repair With In Situ nEedle feNestration of Left Subclavian Artery to Treat AoRtic Dissection(RISEN STAR):A Multicenter Prospective Trial.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IIT20210205B
Record Dates: First submitted 2021-12-27; First posted 2022-01-11 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Aortic Dissection; Left Subclavian Artery Occlusion; Vascular Diseases; Interventional Therapy
MeSH Terms: conditions — Aortic Dissection; Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group RISEN STAR: Patients with Stanford B-type aortic dissection will be treated with endovascular repair with in situ needle fenestration of left subclavian artery.
  Interventions: Behavioral: In situ fenestration

INTERVENTIONS:
Behavioral: In situ fenestration — Interventional therapy of aortic dissection. In situ needle fenestration of left subclavian artery.

SUMMARY:
Background: Aortic dissection (AD) is a common emergency in vascular surgery, which seriously threatens human life and health. The rupture of Stanford type B dissection is located in aortic arch and the dissection range is from the descending aorta or involves the abdominal aorta. At present, the endovascular repair of the thoracic aorta (TEVAR) for AD has been widely deployed worldwide and has become the standard surgical procedure for the treatment of AD. However, there is still controversy regarding the Stanford B aortic dissection that involves the left subclavian artery or the stent landing area less than 1.5 cm.

Study objective: To evaluate the effectiveness and safety of endovascular repair with in situ needle fenestration of left subclavian artery.

Methods: This study intends to enroll 217 patients with Stanford type B aortic dissection who meet the enrollment criteria. The patients will be followed up at 1, 6, 12, and 24 months after endovascular repair, and the CTA images of the thoracic aorta were collected.

ELIGIBILITY:
Inclusion Criteria:

* Based on Computed Tomography Angiography, it is clearly diagnosed as Stanford B type aortic dissection with a breach close to the left subclavian artery;
* The dissection the left subclavian artery, and the proximal landing area is less than 1.5cm. The proximal end of the stent needs to be anchored in zone 2 and the left subclavian needs to be performed arterial revascularization;
* Landing area requirements: no dissection, no intermural hematoma, no severe calcification, no aneurysm-like expansion, diameter 21-44mm, distance between left common carotid artery and left subclavian artery≥10mm;
* The puncture in situ fenestration technique was used to reconstruct the left subclavian artery;
* Signed informed consent;
* Age ≥18 years old, ≤85 years old, no gender limit.

Exclusion Criteria:

* Combined ascending aorta disease or performed ascending aorta surgery before;
* Congenital connective tissue disease (Marfan syndrome, etc.);
* Patients with renal failure or chronic kidney disease before endovascular repair(eGFR≤30ml/min, Dialysis needed, serum creatinine ≥2.5mg/mL within 30 days before operation);
* Cerebral hemorrhage, symptomatic cerebral infarction within 6 weeks before treatment, myocardial infarction within 6 weeks before treatment;
* Combined systemic diseases that cannot be controlled by current medical level (Such as severe heart function, lung function or liver function abnormalities, patients with advanced tumors, patients with cachexia, severe coronary heart disease symptoms that cannot be relieved, abnormal blood coagulation caused by genetic diseases, etc.) ；
* Patient under 18 years or older than 85 years;
* The life expectancy of the patient is shorter than 2 years;
* Those suffering from mental illness or subjectively unable to cooperate;
* Women who are breastfeeding or pregnant, or women or men who have recently had a childbirth plan;
* Currently participating in other interventions research or patients who have been enrolled in this study;
* Have a history of aortic or left subclavian artery surgery;
* Active systemic infection or uncontrolled coagulation dysfunction within 14 days before treatment;
* Those who are unable to take the medication as required by the protocol, or are allergic to antiplatelet drugs (aspirin or clopidogrel), low molecular weight heparin or contrast agents;
* Type II heparin-induced thrombocytopenia (HIT-2) or known hypersensitivity to heparin;
* Thoracic aortic aneurysm, pseudoaneurysm, simple thoracic aortic transmural ulcer, thoracic aortic intermural hematoma;
* There are prominent or irregular thrombus and/or atheroma in the aortic arch or ascending aorta;
* The iliac artery or femoral artery approach is severely diseased and the stent cannot be passed;
* The left subclavian artery is occluded or left Those who have no suitable access for the upper extremities;
* The left subclavian artery is abnormally twisted or angled and is not suitable for fenestration;
* Other conditions that the investigator judges are not suitable for enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Stanford B-type aortic dissection, the proximal landing area is less than 15mm, and the left subclavian artery needs to be reconstructed.
Sampling Method: Non-Probability Sample
Enrollment: 217 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patency rate of main and branch stent. | 1 month after interventional therapy.
  Patency of main and branch stent will be evaluated by Computed Tomography Angiography.
Patency rate of main and branch stent. | 6 months after interventional therapy.
  Patency of main and branch stent will be evaluated by Computed Tomography Angiography.
Patency rate of main and branch stent. | 12 months after interventional therapy
  Patency of main and branch stent will be evaluated by Computed Tomography Angiography.
Patency rate of main and branch stent. | 24 months after interventional therapy
  Patency of main and branch stent will be evaluated by Computed Tomography Angiography.

CONTACTS AND LOCATIONS:
Overall Officials: Hongkun Zhang, Doctor, Study Chair — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eggebrecht H, Mehta RH, Dechene A, Tsagakis K, Kuhl H, Huptas S, Gerken G, Jakob HG, Erbel R. Aortoesophageal fistula after thoracic aortic stent-graft placement: a rare but catastrophic complication of a novel emerging technique. JACC Cardiovasc Interv. 2009 Jun;2(6):570-6. doi: 10.1016/j.jcin.2009.03.010. PMID 19539264
- [Result] Dake MD, Kato N, Mitchell RS, Semba CP, Razavi MK, Shimono T, Hirano T, Takeda K, Yada I, Miller DC. Endovascular stent-graft placement for the treatment of acute aortic dissection. N Engl J Med. 1999 May 20;340(20):1546-52. doi: 10.1056/NEJM199905203402004. PMID 10332016
- [Result] Cambria RP, Conrad MF, Matsumoto AH, Fillinger M, Pochettino A, Carvalho S, Patel V, Matsumura J. Multicenter clinical trial of the conformable stent graft for the treatment of acute, complicated type B dissection. J Vasc Surg. 2015 Aug;62(2):271-8. doi: 10.1016/j.jvs.2015.03.026. PMID 26211376
- [Result] Canaud L, Morishita K, Gandet T, Sfeir J, Bommart S, Alric P, Mandelli M. Homemade fenestrated stent-graft for thoracic endovascular aortic repair of zone 2 aortic lesions. J Thorac Cardiovasc Surg. 2018 Feb;155(2):488-493. doi: 10.1016/j.jtcvs.2017.07.045. Epub 2017 Aug 5. PMID 28867380
- [Result] Xiang Y, Qiu C, He Y, Li D, Shang T, Wu Z, Zhang H. A Single Center Experience of In Situ Needle Fenestration of Supra-aortic Branches During Thoracic Endovascular Aortic Repair. Ann Vasc Surg. 2019 Nov;61:107-115. doi: 10.1016/j.avsg.2019.03.016. Epub 2019 Jun 11. PMID 31200061